CLINICAL TRIAL: NCT01044238
Title: Sustained-Release Methylphenidate for Management of Methamphetamine Dependence
Brief Title: Methylphenidate to Treat Methamphetamine Dependence
Acronym: MPH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Walter Ling, PI, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DA025084 (NIH)
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Methamphetamine Dependence
Keywords: methamphetamine; methylphenidate; clinical trial; random assignment; double blind; abstinence; reduction in methamphetamine use
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active medication (methylphenidate) (Experimental): Condition receiving active medication: 18mg/day during week 1; 36mg/day during week 2; 54mg/day during remainder of study
  Interventions: Drug: methylphenidate
- Placebo (Placebo Comparator): Condition randomly assigned to receive placebo, provided to appear identical to active medication
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: methylphenidate — 18mg/day in week 1; 36mg/day in week 2; 54mg/day in week 3 - participants randomized to either active medication (methylphenidate) or placebo matched to active drug
  Other Names: Concerta
  Arms: active medication (methylphenidate)
Drug: Methylphenidate — 18mg/day for week 1; 36mg/day for week 2; 54mg/day for remainder of study - participants randomized to either active medication (methylphenidate) or placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This 4-year study will investigate the effectiveness of methylphenidate for initiating and sustaining abstinence in methamphetamine dependent individuals. Approximately 90 participants seeking treatment for methamphetamine dependence will be enrolled in the study for an initial 2 weeks to establish clinic compliance. During this compliance phase, participants will receive incentives for clinic attendance. After meeting clinic attendance requirements, participants will be randomized to placebo (n = 45) or active study medication (n = 45) conditions, and given 18mg/daily of study drug or placebo for one week, followed by 36mg/daily study drug/placebo for a second week. Finally, participants will be stabilized on 54mg/daily study drug/placebo for the remainder of the study. Placebo participants will be given placebo medications prepared to appear identical to the active medication. In addition, after randomization, all participants will receive motivational incentives for methamphetamine-negative urine tests and begin weekly cognitive behavioral therapy (CBT) provided for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be seeking treatment for their MA use disorder;
2. Be between 18-55 years of age;
3. Meet DSM-IV-TR criteria for MA dependence as assessed by the Mini International Neuropsychological Interview (MINI);

Exclusion Criteria:

1. Have any history or evidence suggestive of seizures or brain injury;
2. Have any known hypersensitivity or previous medically adverse reaction to methylphenidate;
3. Have a neurological or psychiatric disorder, such as psychosis, bipolar illness, motor tics, Tourette's syndrome, or major depression; organic brain disease or dementia; marked anxiety, tension and agitation; or any psychiatric disorder that would require ongoing treatment or that would make study compliance difficult;
4. Have evidence of clinically significant heart disease or hypertension as determined by medical history or physical examination, including pre-existing heart failure, recent myocardial infarction, ventricular arrhythmia, cardiomyopathy, serious heart rhythm abnormalities, and coronary artery disease.
5. Have a family history in first-degree relatives of early cardiovascular morbidity or mortality, as determined by medical history;
6. Have evidence of an untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease (other than HIV);
7. Have clinically significant abnormal vital signs;
8. Have clinically significant abnormal hematology or chemistry laboratory tests [e.g. liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase), kidney function tests (creatinine and BUN)];
9. Have a baseline ECG that demonstrates clinically significant abnormalities;
10. Have known preexisting severe gastrointestinal narrowing,
11. Be pregnant or nursing. Females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or use a reliable form of contraception including hormonal (oral, Depo-Provera or Nuva-ring), intra-uterine devise, sterilization or double barrier method (simultaneous use of two barrier methods such as condom, diaphragm, spermicide);
12. A history of glaucoma;
13. Use of some medications such as Clonidine, coumarin anticoagulants, anticonvulsants (Phenobarbital, phenytoin, primidone), vasopressor agents, and some antidepressants (tricyclics and selective serotonin reuptake inhibitors),. Also, current use of an MAO inhibitor, or use within 14 days of enrollment;
14. Have any other medical condition that would, in the opinion of the study physician, make participation difficult or unsafe.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
percentage of methamphetamine-negative urine samples compared across two conditions | 14-week study duration

SECONDARY OUTCOMES:
Retention: number of days retained in treatment from randomization to the last scheduled clinic visit | 14 week study duration

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — UCLA Integrated Substance Abuse Programs; Maureen Hillhouse, Ph.D., Study Director — UCLA Integrated Substance Abuse Programs
Locations (1):
- UCLA Integrated Substance Abuse Programs Outpatient Clinical Research Center, Los Angeles, California, United States